CLINICAL TRIAL: NCT00965367
Title: Can Acustimulation Attenuate Postoperative Nausea and Vomiting in Children Who Have Undergone Tonsillectomy/Adenoidectomy?
Brief Title: Postoperative Nausea and Vomiting and Acupuncture/Acupressure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Research Centre of Complementary and Alternative Medicine, Norway (Other)
Collaborators: Lovisenberg Diaconale Hospital (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 125/2007
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Postoperative Vomiting; Nausea
Keywords: POV tonsillectomy adenoidectomy acupuncture acupressure child; Effectiveness of acupuncture on
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acustimulation (Experimental)
  Interventions: Device: Acustimulation
- Standard treatment group (No Intervention)
  Interventions: Device: Acustimulation

INTERVENTIONS:
Device: Acustimulation — Acupressure in P6 bilaterally given after induction of anaesthesia for 20 minutes, followed by acupressure wrist bands applied on the same acupoints for 24 hours.

SUMMARY:
Postoperative nausea and vomiting (PONV) remain a significant challenge in the investigators practice. However, pharmaceutical prophylaxis can imply unpleasant adverse effects. It would therefore be appropriate to consider the use of non-pharmacological methods in preventing PONV. Acupuncture and acupressure are reported to be effective preventive treatment for PONV, and the adverse effects are minimal.

Consequently, the investigators will investigate if acupuncture and acupressure can be implemented as a supplementary to the ordinary treatment in children undergoing surgery for tonsillectomy and/or adenoidectomy. The study will also focus on the feasibility for acupuncture and acupressure in the operation theatre. The study and inclusion/exclusion decisions are conducted after the "intention-to-treat" principle. 126 patients are included, divided into two groups:

1. Treatment Group - standard treatment and acupuncture performed after induction of anaesthesia, acupressure administered before awakening
2. Control Group - standard treatment

The primarily endpoints in this study are nausea, retching and vomiting. The effect of acupuncture/acupressure will be studied with regard to any association with possible factors of predisposition to PONV, as well as with other factors registered during the study. Adverse effects from the acupuncture site and wristband will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for tonsillectomy and/or adenoidectomy
* Informed consent from the parents/guardians

Exclusion Criteria:

* ASA grade greater than or equal to III (patients with severe systemic disease)
* Rash or local infection over an acupuncture point
* Emesis during the previous 24 hours
* Use of medication with antiemetic effect and/or other antiemetic therapy within the 24 hours before surgery
* Gastric or intestinal diseases

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | 24 hours

SECONDARY OUTCOMES:
The effect of the intervention will be studied with regard to any association with possible factors of predisposition to PONV. Adverse effects will also be registered. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arne Johan Norheim, MD Doctor phD, Principal Investigator — National Research Centre of Complementary and Alternative Medicine, Norway
Locations (1):
- Lovisenberg Diaconale Hospital, Oslo, Norway